CLINICAL TRIAL: NCT05137535
Title: A Study of the Infection and Transmission of SARS-CoV-2 in Paediatric Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Collaborators: Azienda ULSS 5 Polesana (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, BRAZZALE ALESSANDRA ROSALBA, Professor, University of Padova
Other Study IDs: PLS COVID 19 - Prog. 3401CESC
Record Dates: First submitted 2021-11-24; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Covid19
Keywords: Covid-19; SARS-CoV-2; children; pediatric; transmission; clinical features
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children diagnosed with Covid-19: Pediatric patients enrolled by the family pediatricians participating in this study, affected by Covid-19 disease whose diagnosis was confirmed by SARS-Cov-2 molecular test
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Family-based questionnaire

SUMMARY:
Covid-19 disease, originated by SARS-Cov-2 Coronavirus, officially appeared in Italy in February 2020. Children and adolescents, in most cases, have an asymptomatic or paucisymptomatic clinical picture and are very rarely hospitalized. Precisely because of the modest symptoms presented, information on the natural history of Covid19 disease and its symptomatology is still limited.

Because almost all children with Covid19 are treated by community medicine, family pediatricians are the most suitable figures to collect the clinical history of these patients.

Information regarding the mode of infection and spread at both the intrafamily and school levels is also poor, and the role that the opening of schools may have on the spread of infection is not yet well established. However, scientific evidence supports the adverse effect of school closures on the physical and mental health of children and adolescents.

Analysis of school spread in a specific area can therefore contribute to increased knowledge about the role of schools, and such information may be useful in guiding health policy choices.

DETAILED DESCRIPTION:
Covid-19 disease, caused by the coronavirus Sars-Cov-2, officially appeared in Italy in February 2020. As of January 2020, the first pediatric cases had already been described, initially in China and then in other countries. Clinical studies suggest that children are susceptible at any age and can transmit the SARS-CoV-2 virus; for the most part pediatric studies analyzed hospitalized patients.

Mainly children and young people present asymptomatic or paucisymptomatic symptoms, and very rarely require hospitalization: the biological reasons for this different clinical picture compared to the adult population are not clear. Just because of the modest symptomatology presented in pediatric age, the natural history of Covid-19 disease and its clinical features in pediatric age are not well known and the disease may be underdiagnosed. Equally scarce is information about Covid-19 spread both within the family and in school communities. These data depend on the availability of tests for the identification of Sars-CoV-2 infection and on how population screenings are organized.

However, knowledge about clinical aspects and diffusion of Covid-19 within the family and at school are fundamental to orient health policy choices such as the opening of schools and of social, educational and sports spaces for children and young people. It is known that transmission of SARS-CoV-2 can occur in school settings, but there are still no definitive data on the impact that this transmission may have on the spread of the infection within the population, because school closures always coincide with closures of other activities and often with general restrictions on the movement of people. Several studies suggest that transmission of SARS-CoV-2 at school is not frequent. School contributes a modest number to the total number of cases and in many cases the infection is attributable to the school staff. Also, the presence of multiple cases in the same school may depend on a greater spread of the virus in the community.

Scientific evidence confirms adverse effect of school closures on the physical and mental health of children and young people, with a very high cost considering impact on learning and reduction of skills in the long term: any reduction in school hours has negative effects on students' cognitive abilities, on the probability of dropping out of school, on college enrollment, and on employment outcomes. In addition, distance learning has exacerbated inequality, because access to computers and the internet is much more complicated for lower class families. Moreover, in some contexts, school closure has generated increases in domestic violence and situations of toxic prolonged stress for children.

The network of community medicine, formed by family pediatricians, represents a unique resource to study Covid-19 natural history in children and spread of disease in their family and at school within a specific territory.

ELIGIBILITY:
Pediatric patients affected by Covid-19 disease whose diagnosis was confirmed by SARS-Cov-2 molecular test enrolled by the family pediatricians participating in this study from February 1 2020 to December 31 2021

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients enrolled by the family pediatricians participating in this study, affected by Covid-19 disease whose diagnosis was confirmed by SARS-Cov-2 molecular test
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Natural history | Feb. 1, 2020 - Dec. 31, 2021
  Description of the natural history of Covid19 in paediatric patients in terms of length, severity and symptoms
Infection and spread | Feb. 1, 2020 - Dec. 31, 2021
  Description of the mode of infection and spread at both the intrafamily and school levels using suitable statistical models

SECONDARY OUTCOMES:
School opening | Feb. 1, 2020 - Dec. 31, 2021
  Study of the impact of school opening on the infection spread using suitable statistical models
Monitoring | Feb. 1, 2020 - Dec. 31, 2021
  Development of a monitoring tool of the spread of infection at school level using GIS technology

CONTACTS AND LOCATIONS:
Locations (1):
- AULSS 5 Polesana, Rovigo, RO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta NS, Mytton OT, Mullins EWS, Fowler TA, Falconer CL, Murphy OB, Langenberg C, Jayatunga WJP, Eddy DH, Nguyen-Van-Tam JS. SARS-CoV-2 (COVID-19): What Do We Know About Children? A Systematic Review. Clin Infect Dis. 2020 Dec 3;71(9):2469-2479. doi: 10.1093/cid/ciaa556. PMID 32392337
- [Background] Posfay-Barbe KM, Wagner N, Gauthey M, Moussaoui D, Loevy N, Diana A, L'Huillier AG. COVID-19 in Children and the Dynamics of Infection in Families. Pediatrics. 2020 Aug;146(2):e20201576. doi: 10.1542/peds.2020-1576. Epub 2020 May 26. No abstract available. PMID 32457213
- [Background] Dorigatti I, Lavezzo E, Manuto L, Ciavarella C, Pacenti M, Boldrin C, Cattai M, Saluzzo F, Franchin E, Del Vecchio C, Caldart F, Castelli G, Nicoletti M, Nieddu E, Salvadoretti E, Labella B, Fava L, Guglielmo S, Fascina M, Grazioli M, Alvisi G, Vanuzzo MC, Zupo T, Calandrin R, Lisi V, Rossi L, Castagliuolo I, Merigliano S, Unwin HJT, Plebani M, Padoan A, Brazzale AR, Toppo S, Ferguson NM, Donnelly CA, Crisanti A. SARS-CoV-2 antibody dynamics and transmission from community-wide serological testing in the Italian municipality of Vo'. Nat Commun. 2021 Jul 19;12(1):4383. doi: 10.1038/s41467-021-24622-7. PMID 34282139
- [Background] European Centre for Disease Prevention and Control. TECHNICAL REPORT COVID-19 in children and the role of school settings in transmission - update 23 December 2020.